CLINICAL TRIAL: NCT03335254
Title: A Phase 1/2a Study to Determine the Dose Response Pharmacokinetics of TSX-011 (Testosterone Undecanoate) in Hypogonadal Males
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Incomplete effect
Sponsor: TesoRx Pharma, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TT-018
Record Dates: First submitted 2017-10-13; First posted 2017-11-07 (Actual); Results first posted 2019-05-16 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-04

CONDITIONS: Hypogonadism; Hypogonadism, Male; Gonadal Disorders; Endocrine System Diseases; Testosterone Deficiency
Keywords: Hypogonadism; Testosterone; Testosterone undecanoate
MeSH Terms: conditions — Hypogonadism; Eunuchism; Gonadal Disorders; Endocrine System Diseases

STUDY DESIGN:
Intervention Model Description: Participants receive identical dosing for Period 1 and Period 2. Beginning with Period 3 subjects are assigned to one of several doses based on dose adjustments. Period 3 dosing groups are run in parallel for the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (20):
- Dose-Escalating Arm 1 (Experimental): Period 1: Single Dose Ascending single-dose period: 190 mg TSX-011 (fed and fasted), 380 mg TSX-011 (fed), and 570 mg TSX-011 (fed).
  Period 2: Twice Daily Dose 380 mg TSX-011 twice daily dosing period of 15 days in fed conditions. Period 3, Day 16-25: Twice Daily Dose If Period 2 Day 8 total testosterone is <350 ng/dL, adjust dose to 570 mg (TU) TSX-011 twice daily.
  Period 3, Day 26-30: Thrice Daily Dose If Period 3 Day 19 total testosterone is <350 ng/dL, dose adjust subjects to 570 mg TSX-011 (TU) dosing thrice daily.
  Assigned Intervention: TSX-011 are capsules with Testosterone Undecanoate (prodrug for androgen testosterone) as the primary ingredient.
  Interventions: Drug: TSX-011
- Dose-Escalating Arm 2 (Experimental): Period 1: Single Dose Ascending single-dose period: 190 mg TSX-011 (fed and fasted), 380 mg TSX-011 (fed), and 570 mg TSX-011 (fed).
  Period 2: Twice Daily Dose 380 mg TSX-011 twice daily dosing period of 15 days in fed conditions. Period 3, Day 16-25: Twice Daily Dose If Period 2 Day 8 total testosterone is <350 ng/dL, adjust dose to 570 mg (TU) TSX-011 twice daily.
  Period 3, Day 26-30: Twice Daily Dose If Period 3 Day 19 total testosterone is ≥350 ng/dL and <500 ng/dL, adjust dose to 633 mg TU twice daily.
  TSX-011: TSX-011 are capsules with Testosterone Undecanoate (prodrug for androgen testosterone) as the primary ingredient.
  Interventions: Drug: TSX-011
- Dose-Escalating Arm 3 (Experimental): Period 1: Single Dose Ascending single-dose period: 190 mg TSX-011 (fed and fasted), 380 mg TSX-011 (fed), and 570 mg TSX-011 (fed).
  Period 2: Twice Daily Dose 380 mg TSX-011 twice daily dosing period of 15 days in fed conditions. Period 3, Day 16-25: Twice Daily Dose If Period 2 Day 8 total testosterone is <350 ng/dL, adjust dose to 570 mg (TU) TSX-011 twice daily.
  Period 3, Day 26-30: Twice Daily Dose If Period 3 Day 19 total testosterone is 500 to 800 ng/dL inclusive, continue current dose 570 mg (TU) TSX-011 twice daily.
  TSX-011: TSX-011 are capsules with Testosterone Undecanoate (prodrug for androgen testosterone) as the primary ingredient.
  Interventions: Drug: TSX-011
- Dose-Escalating Arm 4 (Experimental): Period 1: Single Dose Ascending single-dose period: 190 mg TSX-011 (fed and fasted), 380 mg TSX-011 (fed), and 570 mg TSX-011 (fed).
  Period 2: Twice Daily Dose 380 mg TSX-011 twice daily dosing period of 15 days in fed conditions. Period 3, Day 16-25: Twice Daily Dose If Period 2 Day 8 total testosterone is <350 ng/dL, adjust dose to 570 mg (TU) TSX-011 twice daily.
  Period 3, Day 26-30: Twice Daily Dose If Period 3 Day 19 total testosterone is >800 ng/dL, decrease to 507 mg TU twice daily.
  TSX-011: TSX-011 are capsules with Testosterone Undecanoate (prodrug for androgen testosterone) as the primary ingredient.
  Interventions: Drug: TSX-011
- Dose-Escalating Arm 5 (Experimental): Period 1: Single Dose Ascending single-dose period: 190 mg TSX-011 (fed and fasted), 380 mg TSX-011 (fed), and 570 mg TSX-011 (fed).
  Period 2: Twice Daily Dose 380 mg TSX-011 twice daily dosing period of 15 days in fed conditions. Period 3, Day 16-25: Twice Daily Dose If Period 2 Day 8 total testosterone is ≥350 ng/dL and <500 ng/dL, adjust dose to 443 mg (TU) TSX-011 twice daily.
  Period 3, Day 26-30: Thrice Daily Dose If Period 3 Day 19 total testosterone is <350 ng/dL, dose adjust subjects to 570 mg TSX-011 (TU) dosing thrice daily.
  TSX-011: TSX-011 are capsules with Testosterone Undecanoate (prodrug for androgen testosterone) as the primary ingredient.
  Interventions: Drug: TSX-011
- Dose-Escalating Arm 6 (Experimental): Period 1: Single Dose Ascending single-dose period: 190 mg TSX-011 (fed and fasted), 380 mg TSX-011 (fed), and 570 mg TSX-011 (fed).
  Period 2: Twice Daily Dose 380 mg TSX-011 twice daily dosing period of 15 days in fed conditions. Period 3, Day 16-25: Twice Daily Dose If Period 2 Day 8 total testosterone is ≥350 ng/dL and <500 ng/dL, adjust dose to 443 mg (TU) TSX-011 twice daily.
  Period 3, Day 26-30: Twice Daily Dose If Period 3 Day 19 total testosterone is ≥350 ng/dL and <500 ng/dL, adjust dose to 507 mg TU twice daily.
  TSX-011: TSX-011 are capsules with Testosterone Undecanoate (prodrug for androgen testosterone) as the primary ingredient.
  Interventions: Drug: TSX-011
- Dose-Escalating Arm 7 (Experimental): Period 1: Single Dose Ascending single-dose period: 190 mg TSX-011 (fed and fasted), 380 mg TSX-011 (fed), and 570 mg TSX-011 (fed).
  Period 2: Twice Daily Dose 380 mg TSX-011 twice daily dosing period of 15 days in fed conditions. Period 3, Day 16-25: Twice Daily Dose If Period 2 Day 8 total testosterone is ≥350 ng/dL and <500 ng/dL, adjust dose to 443 mg (TU) TSX-011 twice daily.
  Period 3, Day 26-30: Twice Daily Dose If Period 3 Day 19 total testosterone is 500 to 800 ng/dL inclusive, continue current dose 443 mg (TU) TSX-011 twice daily.
  TSX-011: TSX-011 are capsules with Testosterone Undecanoate (prodrug for androgen testosterone) as the primary ingredient.
  Interventions: Drug: TSX-011
- Dose-Escalating Arm 8 (Experimental): Period 1: Single Dose Ascending single-dose period: 190 mg TSX-011 (fed and fasted), 380 mg TSX-011 (fed), and 570 mg TSX-011 (fed).
  Period 2: Twice Daily Dose 380 mg TSX-011 twice daily dosing period of 15 days in fed conditions. Period 3, Day 16-25: Twice Daily Dose If Period 2 Day 8 total testosterone is ≥350 ng/dL and <500 ng/dL, adjust dose to 443 mg (TU) TSX-011 twice daily.
  Period 3, Day 26-30: Twice Daily Dose If Period 3 Day 19 total testosterone is >800 ng/dL, decrease dose to 380 mg TU twice daily.
  TSX-011: TSX-011 are capsules with Testosterone Undecanoate (prodrug for androgen testosterone) as the primary ingredient.
  Interventions: Drug: TSX-011
- Dose-Escalating Arm 9 (Experimental): Period 1: Single Dose Ascending single-dose period: 190 mg TSX-011 (fed and fasted), 380 mg TSX-011 (fed), and 570 mg TSX-011 (fed).
  Period 2: Twice Daily Dose 380 mg TSX-011 twice daily dosing period of 15 days in fed conditions. Period 3, Day 16-25: Twice Daily Dose If Period 2 Day 8 total testosterone is 500 to 800 ng/dL, inclusive, maintain 380 mg (TU) TSX-011 twice daily.
  Period 3, Day 26-30: Thrice Daily Dose If Period 3 Day 19 total testosterone is <350 ng/dL, dose adjust subjects to 570 mg TSX-011 (TU) dosing thrice daily.
  TSX-011: TSX-011 are capsules with Testosterone Undecanoate (prodrug for androgen testosterone) as the primary ingredient.
  Interventions: Drug: TSX-011
- Dose-Escalating Arm 10 (Experimental): Period 1: Single Dose Ascending single-dose period: 190 mg TSX-011 (fed and fasted), 380 mg TSX-011 (fed), and 570 mg TSX-011 (fed).
  Period 2: Twice Daily Dose 380 mg TSX-011 twice daily dosing period of 15 days in fed conditions. Period 3, Day 16-25: Twice Daily Dose If Period 2 Day 8 total testosterone is 500 to 800 ng/dL, inclusive, maintain 380 mg (TU) TSX-011 twice daily.
  Period 3, Day 26-30: Twice Daily Dose If Period 3 Day 19 total testosterone is ≥350 ng/dL and <500 ng/dL, increase dose to 443 mg TU twice daily.
  TSX-011: TSX-011 are capsules with Testosterone Undecanoate (prodrug for androgen testosterone) as the primary ingredient.
  Interventions: Drug: TSX-011
- Dose-Escalating Arm 11 (Experimental): Period 1: Single Dose Ascending single-dose period: 190 mg TSX-011 (fed and fasted), 380 mg TSX-011 (fed), and 570 mg TSX-011 (fed).
  Period 2: Twice Daily Dose 380 mg TSX-011 twice daily dosing period of 15 days in fed conditions. Period 3, Day 16-25: Twice Daily Dose If Period 2 Day 8 total testosterone is 500 to 800 ng/dL, inclusive, maintain 380 mg (TU) TSX-011 twice daily.
  Period 3, Day 26-30: Twice Daily Dose If Period 3 Day 19 total testosterone is 500 to 800 ng/dL inclusive, continue current dose 380 mg (TU) TSX-011 twice daily.
  TSX-011: TSX-011 are capsules with Testosterone Undecanoate (prodrug for androgen testosterone) as the primary ingredient.
  Interventions: Drug: TSX-011
- Dose-Escalating Arm 12 (Experimental): Period 1: Single Dose Ascending single-dose period: 190 mg TSX-011 (fed and fasted), 380 mg TSX-011 (fed), and 570 mg TSX-011 (fed).
  Period 2: Twice Daily Dose 380 mg TSX-011 twice daily dosing period of 15 days in fed conditions. Period 3, Day 16-25: Twice Daily Dose If Period 2 Day 8 total testosterone is 500 to 800 ng/dL, inclusive, maintain 380 mg (TU) TSX-011 twice daily.
  Period 3, Day 26-30: Twice Daily Dose If Period 3 Day 19 total testosterone is >800 ng/dL, decrease TSX-011 dose to 317 mg TU twice daily.
  TSX-011: TSX-011 are capsules with Testosterone Undecanoate (prodrug for androgen testosterone) as the primary ingredient.
  Interventions: Drug: TSX-011
- Dose-Escalating Arm 13 (Experimental): Period 1: Single Dose Ascending single-dose period: 190 mg TSX-011 (fed and fasted), 380 mg TSX-011 (fed), and 570 mg TSX-011 (fed).
  Period 2: Twice Daily Dose 380 mg TSX-011 twice daily dosing period of 15 days in fed conditions. Period 3, Day 16-25: Twice Daily Dose If Period 2 Day 8 total testosterone is >800 ng/dL, randomize half subjects to receive 317 mg (TU) TSX-011 twice daily Period 3, Day 26-30: Thrice Daily Dose If Period 3 Day 19 total testosterone is <350 ng/dL, dose adjust subjects to 570 mg TSX-011 (TU) dosing thrice daily.
  TSX-011: TSX-011 are capsules with Testosterone Undecanoate (prodrug for androgen testosterone) as the primary ingredient.
  Interventions: Drug: TSX-011
- Dose-Escalating Arm 14 (Experimental): Period 1: Single Dose Ascending single-dose period: 190 mg TSX-011 (fed and fasted), 380 mg TSX-011 (fed), and 570 mg TSX-011 (fed).
  Period 2: Twice Daily Dose 380 mg TSX-011 twice daily dosing period of 15 days in fed conditions. Period 3, Day 16-25: Twice Daily Dose If Period 2 Day 8 total testosterone is >800 ng/dL, randomize half subjects to receive 317 mg (TU) TSX-011 twice daily.
  Period 3, Day 26-30: Twice Daily Dose If Period 3 Day 19 total testosterone is ≥350 ng/dL and <500 ng/dL, increase dose to 380 mg TU twice daily.
  TSX-011: TSX-011 are capsules with Testosterone Undecanoate (prodrug for androgen testosterone) as the primary ingredient.
  Interventions: Drug: TSX-011
- Dose-Escalating Arm 15 (Experimental): Period 1: Single Dose Ascending single-dose period: 190 mg TSX-011 (fed and fasted), 380 mg TSX-011 (fed), and 570 mg TSX-011 (fed).
  Period 2: Twice Daily Dose 380 mg TSX-011 twice daily dosing period of 15 days in fed conditions. Period 3, Day 16-25: Twice Daily Dose If Period 2 Day 8 total testosterone is >800 ng/dL, randomize half subjects to receive 317 mg (TU) TSX-011 twice daily.
  Period 3, Day 26-30: Twice Daily Dose If Period 3 Day 19 total testosterone is 500 to 800 ng/dL inclusive, continue current dose 317 mg (TU) TSX-011 twice daily.
  TSX-011: TSX-011 are capsules with Testosterone Undecanoate (prodrug for androgen testosterone) as the primary ingredient.
  Interventions: Drug: TSX-011
- Dose-Escalating Arm 16 (Experimental): Period 1: Single Dose Ascending single-dose period: 190 mg TSX-011 (fed and fasted), 380 mg TSX-011 (fed), and 570 mg TSX-011 (fed).
  Period 2: Twice Daily Dose 380 mg TSX-011 twice daily dosing period of 15 days in fed conditions. Period 3, Day 16-25: Twice Daily Dose If Period 2 Day 8 total testosterone is >800 ng/dL, randomize half subjects to receive 317 mg (TU) TSX-011 twice daily.
  Period 3, Day 26-30: Twice Daily Dose If Period 3 Day 19 total testosterone is >800 ng/dL, decrease dose to 253 mg TU twice daily.
  TSX-011: TSX-011 are capsules with Testosterone Undecanoate (prodrug for androgen testosterone) as the primary ingredient.
  Interventions: Drug: TSX-011
- Dose-Escalating Arm 17 (Experimental): Period 1: Single Dose Ascending single-dose period: 190 mg TSX-011 (fed and fasted), 380 mg TSX-011 (fed), and 570 mg TSX-011 (fed).
  Period 2: Twice Daily Dose 380 mg TSX-011 twice daily dosing period of 15 days in fed conditions. Period 3, Day 16-25: Once Daily Dose If Period 2 Day 8 total testosterone is >800 ng/dL, randomize half subjects to receive 507 mg (TU) TSX-011 once daily.
  Period 3, Day 26-30: Thrice Daily Dose If Period 3 Day 19 total testosterone is <350 ng/dL, dose adjust subjects to 570 mg TSX-011 (TU) dosing thrice daily.
  TSX-011: TSX-011 are capsules with Testosterone Undecanoate (prodrug for androgen testosterone) as the primary ingredient.
  Interventions: Drug: TSX-011
- Dose-Escalating Arm 18 (Experimental): Period 1: Single Dose Ascending single-dose period: 190 mg TSX-011 (fed and fasted), 380 mg TSX-011 (fed), and 570 mg TSX-011 (fed).
  Period 2: Twice Daily Dose 380 mg TSX-011 twice daily dosing period of 15 days in fed conditions. Period 3, Day 16-25: Once Daily Dose If Period 2 Day 8 total testosterone is >800 ng/dL, randomize half subjects to receive 507 mg (TU) TSX-011 once daily.
  Period 3, Day 26-30: Once Daily Dose If Period 3 Day 19 total testosterone is ≥350 ng/dL and <500 ng/dL, dose adjust subjects on once-daily dosing from 507 mg TU daily to 570 mg TU daily.
  TSX-011: TSX-011 are capsules with Testosterone Undecanoate (prodrug for androgen testosterone) as the primary ingredient.
  Interventions: Drug: TSX-011
- Dose-Escalating Arm 19 (Experimental): Period 1: Single Dose Ascending single-dose period: 190 mg TSX-011 (fed and fasted), 380 mg TSX-011 (fed), and 570 mg TSX-011 (fed).
  Period 2: Twice Daily Dose 380 mg TSX-011 twice daily dosing period of 15 days in fed conditions. Period 3, Day 16-25: Once Daily Dose If Period 2 Day 8 total testosterone is >800 ng/dL, randomize half subjects to receive 507 mg (TU) TSX-011 once daily.
  Period 3, Day 26-30: Once Daily Dose If Period 3 Day 19 total testosterone is 500 to 800 ng/dL inclusive, continue current dose of 507 mg TU daily.
  TSX-011: TSX-011 are capsules with Testosterone Undecanoate (prodrug for androgen testosterone) as the primary ingredient.
  Interventions: Drug: TSX-011
- Dose-Escalating Arm 20 (Experimental): Period 1: Single Dose Ascending single-dose period: 190 mg TSX-011 (fed and fasted), 380 mg TSX-011 (fed), and 570 mg TSX-011 (fed).
  Period 2: Twice Daily Dose 380 mg TSX-011 twice daily dosing period of 15 days in fed conditions. Period 3, Day 16-25: Once Daily Dose If Period 2 Day 8 total testosterone is >800 ng/dL, randomize half subjects to receive 507 mg (TU) TSX-011 once daily.
  Period 3, Day 26-30: Once Daily Dose If Period 3, Day 19 total testosterone is >800 ng/dL, decrease dose to 380 mg TU daily.
  TSX-011: TSX-011 are capsules with Testosterone Undecanoate (prodrug for androgen testosterone) as the primary ingredient.
  Interventions: Drug: TSX-011

INTERVENTIONS:
Drug: TSX-011 — TSX-011 are capsules with Testosterone Undecanoate (prodrug for androgen testosterone) as the primary ingredient.

SUMMARY:
This will be a phase 1/2a, open-label, single-center study with 3 periods. The aims of the study are to:

1. evaluate the dose-response curve following ascending single doses of TSX-011;
2. confirm optimum dosing conditions;
3. evaluate the efficacy of single or multiple daily adaptive dosing; and
4. evaluate the safety and tolerability of TSX-011.

DETAILED DESCRIPTION:
This will be a phase 1/2a, open-label, single-center study with 3 periods. The aims of the study are to: 1) evaluate the dose-response curve following ascending single doses of TSX-011; 2) confirm optimum dosing conditions; 3) evaluate the efficacy of single or multiple daily adaptive dosing; and 4) evaluate the safety and tolerability of TSX-011. Up to 24 hypogonadal men will be enrolled in this study to yield 16 evaluable subjects, and it is desired that the same 24 subjects participate in all 3 study periods.

Period 1 is an ascending single-dose study of TSX-011 at 3 doses, with the lowest dose administered under fed and fasted conditions: 190 mg TSX-011 in the fed state, 190 mg TSX-011 in the fasted state, 380 mg TSX-011 in the fed state, and 570 mg TSX-011 in the fed state. Before exposure to TSX-011, a 24 hour baseline measurement of testosterone and DHT will be performed for each subject. Samples for analysis of testosterone will be obtained at the following time points on Day -1: hour 0 (8 am ± 60 minutes) and 1.5, 3, 4.5, 6, 8, 12, 16, and 24 hours (± 15 minutes for each time point).

The day following the sampling for endogenous testosterone (Day 1) in Period 1, each subject will receive the first single dose of TSX-011 (190 mg) under fed conditions. Following administration of TSX-011, blood samples will be obtained over a 24-hour period for PK analysis. Subjects will undergo a minimum 3-day and up to 7-day washout period between each of the doses of TSX-011 in Period 1. After the 570 mg TSX 011 dose in Period 1, a minimum 3-day and up to 7-day washout period will occur before the start of Period 2.

Period 2 is a twice-daily dosing period, where fed subjects will be dosed with 380 mg TSX-011 twice daily for 15 days (Days 1 through 15). Pharmacokinetic assessments over 24 hours will occur on Days 1 and 15. The TSX-011 dose will be titrated up or down beginning with the Day 16 (Period 3) morning dose, based on established dosing rules.

Period 3 is a dose-adjusted adaptive design period that begins on Day 16, with the first adjusted TSX-011 dose administered in the fed state on a once-daily or twice-daily schedule. The 6-hour postdose (± 15 minutes) testosterone level on Day 19 will be used to perform the second and final TSX-011 dose adjustment, based on established criteria. As specified by the dose adjustment rules, Day 26 begins with either a once-daily, twice-daily, or thrice-daily fed dose schedule. The thrice-daily dose schedule will be administered only to non-responders. On Day 30, a 24 hour PK assessment will be performed, and the subject's participation in the study is completed the morning of Day 31.

ELIGIBILITY:
Inclusion Criteria:

* Testosterone level <350 ng/dL, 10 am [± 2 hour] sample.
* Body mass index (BMI) <35.0 kg/m2 and weight ≥50 kg

Exclusion Criteria:

* History of clinically significant renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, psychiatric, or cardiovascular disease or any other condition.
* Significant gastrointestinal or malabsorption conditions.
* Any man in whom testosterone therapy is contraindicated including the following:

  1. Known or suspected carcinoma (or history of carcinoma) of the prostate, clinically significant symptoms of benign prostatic hyperplasia, and/or clinically significant symptoms of lower urinary obstruction and International Prostate Symptom Score (IPSS) ≥19. A clinically significant digital rectal examination of the prostate or clinically significant elevated serum PSA levels (>4.0 ng/mL).
  2. Known or suspected carcinoma (or history of carcinoma) of the breast.
  3. Liver disease defined as alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2 × upper limit of normal (ULN) or bilirubin >2 × ULN.
  4. Active deep vein thrombosis or thromboembolic disorder, or a documented history of these conditions.
  5. Untreated sleep apnea.
  6. Hematocrit >50%.
  7. Untreated moderate to severe depression.
* Current use of long-acting testosterone or any of the testosterone esters injectables.
* Topical, oral, or injectable testosterone replacement therapy.
* Clinically significant changes in any medications (including dosages) or medical conditions in the 28 days before screening.
* Suspected reversible hypogonadism (e.g., leuprolide injection).
* Taking concomitant medications that affect testosterone concentrations or metabolism
* Uncontrolled diabetes (screening glycated hemoglobin [HbA1c] ≥9%).
* Donated blood or blood products or experienced significant blood loss within 90 days before dosing.
* Donated bone marrow within 6 months before dosing.
* History of drug or alcohol abuse in the last 6 months.
* Ingested St John's wort within 30 days of screening.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2018-05-03 (Actual); Study Completion 2018-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Oefelein, MD, Study Director — TesoRx Pharma
Locations (1):
- California Clinical Trials, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial enrolled nine male subjects. All subjects received treatment and completed the study. None of the enrolled/randomized subjects were withdrawn or discontinued from the study.
Groups:
- Dose-Escalating Arm 1: Period 1: Single Dose Ascending single-dose period: 190 mg TSX-011 (fed and fasted), 380 mg TSX-011 (fed), and 570 mg TSX-011 (fed).
  Period 2: Twice Daily Dose 380 mg TSX-011 twice daily dosing period of 15 days in fed conditions. Period 3, Day 16-25: Twice Daily Dose If Period 2 Day 8 total testosterone is <350 ng/dL, adjust dose to 570 mg (TU) TSX-011 twice daily.
  Period 3, Day 26-30: Thrice Daily Dose If Period 3 Day 19 total testosterone is <350 ng/dL, dose adjust subjects to 570 mg TSX-011 (TU) dosing thrice daily.
  TSX-011: TSX-011 are capsules with Testosterone Undecanoate (prodrug for androgen testosterone) as the primary ingredient.
Period: Period 1
Arm/Group | Dose-Escalating Arm 1 | Dose-Escalating Arm 2 | Dose-Escalating Arm 3 | Dose-Escalating Arm 4 | Dose-Escalating Arm 5 | Dose-Escalating Arm 6 | Dose-Escalating Arm 7 | Dose-Escalating Arm 8 | Dose-Escalating Arm 9 | Dose-Escalating Arm 10 | Dose-Escalating Arm 11 | Dose-Escalating Arm 12 | Dose-Escalating Arm 13 | Dose-Escalating Arm 14 | Dose-Escalating Arm 15 | Dose-Escalating Arm 16 | Dose-Escalating Arm 17 | Dose-Escalating Arm 18 | Dose-Escalating Arm 19 | Dose-Escalating Arm 20
Started | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2, Day 1-15
Arm/Group | Dose-Escalating Arm 1 | Dose-Escalating Arm 2 | Dose-Escalating Arm 3 | Dose-Escalating Arm 4 | Dose-Escalating Arm 5 | Dose-Escalating Arm 6 | Dose-Escalating Arm 7 | Dose-Escalating Arm 8 | Dose-Escalating Arm 9 | Dose-Escalating Arm 10 | Dose-Escalating Arm 11 | Dose-Escalating Arm 12 | Dose-Escalating Arm 13 | Dose-Escalating Arm 14 | Dose-Escalating Arm 15 | Dose-Escalating Arm 16 | Dose-Escalating Arm 17 | Dose-Escalating Arm 18 | Dose-Escalating Arm 19 | Dose-Escalating Arm 20
Started | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3, Day 16-25
Arm/Group | Dose-Escalating Arm 1 | Dose-Escalating Arm 2 | Dose-Escalating Arm 3 | Dose-Escalating Arm 4 | Dose-Escalating Arm 5 | Dose-Escalating Arm 6 | Dose-Escalating Arm 7 | Dose-Escalating Arm 8 | Dose-Escalating Arm 9 | Dose-Escalating Arm 10 | Dose-Escalating Arm 11 | Dose-Escalating Arm 12 | Dose-Escalating Arm 13 | Dose-Escalating Arm 14 | Dose-Escalating Arm 15 | Dose-Escalating Arm 16 | Dose-Escalating Arm 17 | Dose-Escalating Arm 18 | Dose-Escalating Arm 19 | Dose-Escalating Arm 20
Started | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3, Day 26-30
Arm/Group | Dose-Escalating Arm 1 | Dose-Escalating Arm 2 | Dose-Escalating Arm 3 | Dose-Escalating Arm 4 | Dose-Escalating Arm 5 | Dose-Escalating Arm 6 | Dose-Escalating Arm 7 | Dose-Escalating Arm 8 | Dose-Escalating Arm 9 | Dose-Escalating Arm 10 | Dose-Escalating Arm 11 | Dose-Escalating Arm 12 | Dose-Escalating Arm 13 | Dose-Escalating Arm 14 | Dose-Escalating Arm 15 | Dose-Escalating Arm 16 | Dose-Escalating Arm 17 | Dose-Escalating Arm 18 | Dose-Escalating Arm 19 | Dose-Escalating Arm 20
Started | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Under the same Period of the trial, only one dosing group was selected based on the adaptive dosing criteria. Therefore, some groups showed zero participants.
Groups:
- Dose-Escalating Arm 1: Period 1: Single Dose Ascending single-dose period: 190 mg TSX-011 (fed and fasted), 380 mg TSX-011 (fed), and 570 mg TSX-011 (fed).
  Period 2: Twice Daily Dos 380 mg TSX-011 twice daily dosing period of 15 days in fed conditions. Period 3, Day 16-25: Twice Daily Dose If Period 2 Day 8 total testosterone is <350 ng/dL, adjust dose to 570 mg (TU) TSX-011 twice daily.
  Period 3, Day 26-30: Thrice Daily Dose If Period 3 Day 19 total testosterone is <350 ng/dL, dose adjust subjects to 570 mg TSX-011 (TU) dosing thrice daily.
  TSX-011: TSX-011 are capsules with Testosterone Undecanoate (prodrug for androgen testosterone) as the primary ingredient.
- Total: Total of all reporting groups
Arm/Group | Dose-Escalating Arm 1 | Dose-Escalating Arm 2 | Dose-Escalating Arm 3 | Dose-Escalating Arm 4 | Dose-Escalating Arm 5 | Dose-Escalating Arm 6 | Dose-Escalating Arm 7 | Dose-Escalating Arm 8 | Dose-Escalating Arm 9 | Dose-Escalating Arm 10 | Dose-Escalating Arm 11 | Dose-Escalating Arm 12 | Dose-Escalating Arm 13 | Dose-Escalating Arm 14 | Dose-Escalating Arm 15 | Dose-Escalating Arm 16 | Dose-Escalating Arm 17 | Dose-Escalating Arm 18 | Dose-Escalating Arm 19 | Dose-Escalating Arm 20 | Total
Number analyzed (Participants) | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 0
  Between 18 and 65 years | 9 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 9
  >=65 years | 0 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 0
Age, Continuous [Mean (Standard Deviation); unit: yr] | 51.9 (6.66) |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 51.9 (6.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 0
  Male | 9 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 0
  Asian | 4 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 4
  Native Hawaiian or Other Pacific Islander | 0 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 0
  Black or African American | 1 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 1
  White | 4 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 4
  More than one race | 0 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 0
  Unknown or Not Reported | 0 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders Based on Measured Total Testosterone (Cavg).
Description: TSX-011 responders are defined as study subjects who are able to achieve a Cavg serum total testosterone > 350 ng/dL. The percentage of responders is recorded for each treatment group within each period.
Time Frame: Period 1: Up to 13 days. Period 2: 15 days. Period 3: 15 days.
Population: Arm 2 to Arm 20 have zero participants due to dose adjustment based on the total testosterone levels presented.
Measure: Number; unit: percentage of participants
Arm/Group | Dose-Escalating Arm 1 | Dose-Escalating Arm 2 | Dose-Escalating Arm 3 | Dose-Escalating Arm 4 | Dose-Escalating Arm 5 | Dose-Escalating Arm 6 | Dose-Escalating Arm 7 | Dose-Escalating Arm 8 | Dose-Escalating Arm 9 | Dose-Escalating Arm 10 | Dose-Escalating Arm 11 | Dose-Escalating Arm 12 | Dose-Escalating Arm 13 | Dose-Escalating Arm 14 | Dose-Escalating Arm 15 | Dose-Escalating Arm 16 | Dose-Escalating Arm 17 | Dose-Escalating Arm 18 | Dose-Escalating Arm 19 | Dose-Escalating Arm 20
Number analyzed (Participants) | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
percentage of participants
  Period 1 | 33.33 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |
  Period 2 | 22.22 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |
  Period 3, Day 15-26 | 0 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |
  Period 3, Day 26-30 | 0 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |

ADVERSE EVENTS:
Time Frame: Adverse events presented were collected from 1 December 2017 (first subject Day 0) and 17 May 2018 (last subject visit).
Description: An adverse event is considered any untoward or unfavorable medical occurrence associated with the subject's participation in the study. Subjects were asked an open question such as "How have you been feeling since you were last asked?" at all visits from Day 0 to Exit.
Groups:
- Period 1: Single Dose: Period 1. Ascending single-dose period: 190 mg TSX-011 (fed and fasted), 380 mg TSX-011 (fed), and 570 mg TSX-011 (fed).
  TSX-011: TSX-011 are capsules with Testosterone Undecanoate (prodrug for androgen testosterone) as the primary ingredient.
- Period 2: Twice Daily Dose: 380 mg TSX-011 twice daily dosing period of 15 days in fed conditions.
  TSX-011: TSX-011 are capsules with Testosterone Undecanoate (prodrug for androgen testosterone) as the primary ingredient.
- Period 3, Day 16-25: Once Daily Dose: If Period 2 Day 8 total testosterone is >800 ng/dL, subjects randomized in a 1:1 ratio to receive:
  * Schedule A: 317 mg (TU) TSX-011 twice daily OR
  * Schedule B: 507 mg (TU) TSX-011 once daily.
  TSX-011: TSX-011 are capsules with Testosterone Undecanoate (prodrug for androgen testosterone) as the primary ingredient.
- Period 3, Day 16-25: Twice Daily Dose: If Period 2 Day 8 total testosterone is <350 ng/dL, adjust dose to 570 mg (TU) TSX-011 twice daily.
  If Period 2 Day 8 total testosterone is ≥350 ng/dL and <500 ng/dL, adjust dose to 443 mg (TU) TSX-011 twice daily.
  If Period 2 Day 8 total testosterone is 500 to 800 ng/dL, inclusive, maintain 380 mg (TU) TSX-011 twice daily.
  If Period 2 Day 8 total testosterone is >800 ng/dL, randomize subjects in a 1:1 ratio to receive:
  * Schedule A: 317 mg (TU) TSX-011 twice daily OR
  * Schedule B: 507 mg (TU) TSX-011 once daily.
  TSX-011: TSX-011 are capsules with Testosterone Undecanoate (prodrug for androgen testosterone) as the primary ingredient.
- Period 3, Day 26-30: Once Daily Dose: If Period 3 Day 19 total testosterone is ≥350 ng/dL and <500 ng/dL:
  Dose adjust subjects on once-daily dosing from 507 mg TU daily to 570 mg TU daily.
  If Period 3 Day 19 total testosterone is 500 to 800 ng/dL inclusive, continue current dose of 507 mg TU daily.
  If Period 3, Day 19 total testosterone is >800 ng/dL, decrease TSX-011 dose as follows: Dose adjust subjects on once-daily dosing from 507 mg TU daily to 380 mg TU daily.
  TSX-011: TSX-011 are capsules with Testosterone Undecanoate (prodrug for androgen testosterone) as the primary ingredient.
- Period 3, Day 26-30: Twice Daily Dose: If Period 3 Day 19 total testosterone is ≥350 ng/dL and <500 ng/dL:
  Dose adjust subjects on twice daily dosing as follows:
  * If dose is 570 mg TU twice daily, increase to 633 mg TU twice daily.
  * If dose is 443 mg TU twice daily, increase to 507 mg TU twice daily.
  * If dose is 380 mg TU twice daily, increase to 443 mg TU twice daily.
  * If dose is 317 mg TU twice daily, increase to 380 mg TU twice daily. If Period 3 Day 19 total testosterone is 500 to 800 ng/dL inclusive, continue current dose twice daily.
  If Period 3 Day 19 total testosterone is >800 ng/dL, decrease TSX-011 dose as follows:
  For the twice-daily dosing group:
  * If dose is 570 mg TU twice daily, decrease to 507 mg TU twice daily.
  * If dose is 443 mg TU twice daily, decrease to 380 mg TU twice daily.
  * If dose is 380 mg TU twice daily, decrease to 317 mg TU twice daily.
  * If dose is 317 mg TU twice daily, decrease to 253 mg TU twice daily. TSX-011 are capsules with primarily Testosterone Undecanoate.
- Period 3, Day 26-30: Thrice Daily Dose: If Period 3 Day 19 total testosterone is <350 ng/dL, dose adjust subjects to 570 mg TSX-011 (TU) dosing thrice daily.
  TSX-011: TSX-011 are capsules with Testosterone Undecanoate (prodrug for androgen testosterone) as the primary ingredient.
Arm/Group | Period 1: Single Dose | Period 2: Twice Daily Dose | Period 3, Day 16-25: Once Daily Dose | Period 3, Day 16-25: Twice Daily Dose | Period 3, Day 26-30: Once Daily Dose | Period 3, Day 26-30: Twice Daily Dose | Period 3, Day 26-30: Thrice Daily Dose
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/0 | 0/9 | 0/0 | 0/0 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/0 | 0/9 | 0/0 | 0/0 | 0/9
Other Adverse Events (participants affected / at risk) | 2/9 | 1/9 | 0/0 | 0/9 | 0/0 | 0/0 | 2/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: Single Dose (N=9) | Period 2: Twice Daily Dose (N=9) | Period 3, Day 16-25: Once Daily Dose (N=0) | Period 3, Day 16-25: Twice Daily Dose (N=9) | Period 3, Day 26-30: Once Daily Dose (N=0) | Period 3, Day 26-30: Twice Daily Dose (N=0) | Period 3, Day 26-30: Thrice Daily Dose (N=9)
Insect Bite/Arthropod Bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lightheaded/Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye Irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever/Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor will review and provide prior written consent, which shall not be unreasonably withheld.

PI will be permitted to publish in journals, theses, dissertations, or other formats of their own choosing.

DOCUMENTS (2):
  • Study Protocol (2018-03-05): https://cdn.clinicaltrials.gov/large-docs/54/NCT03335254/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-13): https://cdn.clinicaltrials.gov/large-docs/54/NCT03335254/SAP_001.pdf